CLINICAL TRIAL: NCT06619353
Title: Residual CardioVascular Risk (RCVR) After Percutaneous Coronary Intervention: a Prospective Multicenter Study
Brief Title: RCVR (Residual CardioVascular Risk) Prospective Multicenter Study
Acronym: RCVR
Status: Recruiting | Type: Observational
Sponsor: CHA University (Other)
Responsible Party: Principal Investigator, Seung-Yul Lee, Associate Professor, CHA University
Other Study IDs: CHAMC IRB 2024-01-054-004
Record Dates: First submitted 2024-09-23; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Coronary Artery Disease
Keywords: Percutaneous Coronary Intervention
MeSH Terms: conditions — Coronary Artery Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Residual CardioVascular Risk: Residual cardiovascular risk is assessed in patients undergoing PCI.
  Interventions: Diagnostic Test: Blood Sample; Other: DICOM Dataset

INTERVENTIONS:
Diagnostic Test: Blood Sample — Patients' blood samples are tested at 1 month, and then annually for 3 years post-intervention to assess residual thrombotic, metabolic, and inflammatory risk.
Other: DICOM Dataset — Patients' DICOM dataset is evaluated using artificial intelligence-based quantitative coronary analysis to assess a procedural risk.

SUMMARY:
The observational study aims to evaluate the long-term effects of residual cardiovascular risk on clinical outcomes following percutaneous coronary intervention (PCI). This risk includes thrombotic, metabolic, inflammatory, and procedural factors, which are assessed 1 month after the intervention. The primary question the study seeks to answer is:

What residual cardiovascular risk affects long-term clinical outcomes in patients undergoing PCI?

Participants will undergo artificial intelligence-based quantitative coronary analysis after PCI and will have comprehensive laboratory tests conducted at 1 month to evaluate residual cardiovascular risk, and then annually for 3 years post-intervention to assess changes in this risk.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone percutaneous coronary intervention.
* Patients who have provided written informed consent.

Exclusion Criteria:

* Under 19 years of age.
* Pregnant, breastfeeding, or women of childbearing age.
* Currently has a malignancy or has a history of malignancy within the past 5 years.
* Life expectancy of less than 5 years.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing PCI
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-06-17 (Actual); Primary Completion 2029-06-17 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Net adverse clinical event | 3 years post-intervention
  The composite of cardiovascular death, nonfatal spontaneous (nonprocedural) myocardial infarction, nonfatal ischemic stroke, unplanned hospitalization leading to urgent revascularization, and major bleeding.

SECONDARY OUTCOMES:
Cardiovascular death | 3 years post-intervention
  The composite of cardiac and vascular death. Any death due to proximate cardiac cause (eg, myocardial infarction, low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause, and all procedure-related deaths, including those related to concomitant treatment, will be classified as cardiac death. Death caused by noncoronary vascular causes, such as cerebrovascular disease, pulmonary embolism, ruptured aortic aneurysm, dissecting aneurysm, or other vascular diseases will be classified as vascular death.
Nonfatal spontaneous (nonprocedural) myocardial infarction | 3 years post-intervention
  Myocardial infarction is defined as symptoms, electrocardiographic changes, or abnormal imaging findings, combined with a creatine kinase MB fraction above the upper normal limits or a troponin T or troponin I level greater than the 99th percentile of the upper normal limit. Myocardial infarction that are not associated with a revascularization procedure will be classified as nonfatal spontaneous myocardial infarction.
Nonfatal ischemic stroke | 3 years post-intervention
  Cerebrovascular event resulting in a neurologic deficit within 24 hours or the presence of acute infarction as demonstrated by imaging studies will be classified as nonfatal ischemic stroke.
Unplanned hospitalization leading to urgent revascularization | 3 years post-intervention
  This event will be present only if the participant is hospitalized unexpectedly because of persisting or increasing complaints of chest pain (with or without ST-T changes, with or without elevated biomarkers) and a revascularization is performed within the same hospitalization. It should be clearly distinguished from the revascularization procedure which is performed on non-urgent basis.
Major bleeding | 3 years post-intervention
  Bleeding Academic Research Consortium type 3 or 5
V-Angiographic success | Within 1 hour post-intervention
  Participant with visually estimated residual diameter stenosis of less than 20% in all PCI-treated lesions
V-Complete revascularization | Within 1 hour post-intervention
  Participant without angiographically significant stenosis (visually estimated diameter stenosis severity of ≥70% for non-left main disease and ≥50% for left main disease) after PCI in entire coronary arteries
AI-Angiographic success | Within 1 hour post-intervention
  Participant with artificial intelligence-measured residual diameter stenosis of less than 20% in all PCI-treated lesions
AI-Complete revascularization | Within 1 hour post-intervention
  Participant without angiographically significant stenosis (artificial intelligence-measured diameter stenosis severity of ≥70% for non-left main disease and ≥50% for left main disease) after PCI in entire coronary arteries
Platelet reactivity | 1 month, 1 year, 2 years, and 3 years post-intervention
  This will be measured with P2Y12 reaction units through VerifyNow test.
Thrombogenicity profiles | 1 month, 1 year, 2 years, and 3 years post-intervention
  This will include R, K, Angle, A10, MA, and Ly30 through thromboelastography.
Lipid profiles | 1 month, 1 year, 2 years, and 3 years post-intervention
  This will include total cholesterol, high-density lipoprotein, low-density lipoprotein, and lipoprotein (a).
Hemoglobin A1C | 1 month, 1 year, 2 years, and 3 years post-intervention
High-sensitivity C-reactive protein | 1 month, 1 year, 2 years, and 3 years post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Yul Lee, MD, Principal Investigator — CHA Bundang Medical Center
Locations (1):
- CHA Bundang Medical Center, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dhindsa DS, Sandesara PB, Shapiro MD, Wong ND. The Evolving Understanding and Approach to Residual Cardiovascular Risk Management. Front Cardiovasc Med. 2020 May 13;7:88. doi: 10.3389/fcvm.2020.00088. eCollection 2020. PMID 32478100
- [Background] Cutlip DE, Windecker S, Mehran R, Boam A, Cohen DJ, van Es GA, Steg PG, Morel MA, Mauri L, Vranckx P, McFadden E, Lansky A, Hamon M, Krucoff MW, Serruys PW; Academic Research Consortium. Clinical end points in coronary stent trials: a case for standardized definitions. Circulation. 2007 May 1;115(17):2344-51. doi: 10.1161/CIRCULATIONAHA.106.685313. PMID 17470709
- [Background] Mehran R, Rao SV, Bhatt DL, Gibson CM, Caixeta A, Eikelboom J, Kaul S, Wiviott SD, Menon V, Nikolsky E, Serebruany V, Valgimigli M, Vranckx P, Taggart D, Sabik JF, Cutlip DE, Krucoff MW, Ohman EM, Steg PG, White H. Standardized bleeding definitions for cardiovascular clinical trials: a consensus report from the Bleeding Academic Research Consortium. Circulation. 2011 Jun 14;123(23):2736-47. doi: 10.1161/CIRCULATIONAHA.110.009449. No abstract available. PMID 21670242